CLINICAL TRIAL: NCT06044948
Title: Clinical Assessment of a Daily Disposable Soft Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLU484-P003
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Refractive Errors
Keywords: Contact Lenses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Masking Description: In this single arm study, the subject will be masked to the lens type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DAILIES TOTAL1 (Experimental): Delefilcon A contact lenses worn in both eyes for the typical number of hours the subject wears his/her habitual contact lenses. The lenses will be worn in a daily disposable manner.
  Interventions: Device: Delefilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses — Daily disposable, silicone hydrogel spherical contact lenses
  Other Names: DAILIES TOTAL1

SUMMARY:
The purpose of this study is to assess the clinical performance of DAILIES TOTAL1® spherical soft contact lenses over approximately 1 week of daily wear.

DETAILED DESCRIPTION:
Subjects will be expected to attend 2 visits (Visit 1 Screen/Baseline/ Dispense; and Visit 2 Week 1 Follow-up/ Exit). The total duration of a subject's participation in the study as well as exposure to the contact lenses will be approximately 1 week (6-8 days of contact lens wear).

ELIGIBILITY:
Key Inclusion Criteria:

* Current wearer of commercial spherical soft contact lenses in both eyes with at least 3 months of wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day;
* Manifest cylinder less than or equal to 0.75 diopter (D) in each eye;
* Best corrected distance visual acuity better than or equal to 20/25 (Snellen) in each eye.

Key Exclusion Criteria:

* Current or prior habitual DAILIES TOTAL1 soft contact lens wear in the past 3 months prior to consent;
* Monovision contact lens wear;
* Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CRD Vision Care, Study Director — Alcon Research, LLC
Locations (6):
- United States (6):
  - Tallahassee Eye Center, Tallahassee, Florida
  - The Eye Doctors, Inc., Eden Prairie, Minnesota
  - Oculus Research, Inc., Garner, North Carolina
  - ProCare Vision Center, Granville, Ohio
  - Wyomissing Optometric Center, Wyomissing, Pennsylvania
  - Optometry Group, PLLC, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 investigative sites located in 1 country (US).
Pre-assignment Details: Of the 97 enrolled, 1 subject was exited as a screen failure prior to being exposed to the product. This reporting group includes all participants who were exposed to the product (96).
Units Other Than Participants: eyes
Groups:
- DAILIES TOTAL1: Delefilcon A contact lenses (daily disposable, silicone hydrogel spherical contact lenses) worn in both eyes for the typical number of hours the subject wears his/her habitual contact lenses. The lenses were worn in a daily disposable manner.
Period: Overall Study
Arm/Group | DAILIES TOTAL1
Started | 96; 192 eyes
Completed | 96; 192 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all subjects/eyes exposed to DAILIES TOTAL1 lenses evaluated in this study.
Arm/Group | DAILIES TOTAL1
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 83
  Black or African American | 9
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Other | 2
  Multi-racial | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 93

OUTCOME MEASURES:

1. Primary Outcome: Distance VA With Study Lenses at Week 1
Description: Visual acuity (VA) was measured for each eye individually with study lenses on eye using letter charts. VA was recorded in Snellen where 20/20 represents normal distance eyesight and 20/15 represents better than normal eyesight. No hypothesis testing was prespecified for this endpoint.
Time Frame: Week 1
Population: The safety analysis set included all subjects/eyes exposed to DAILIES TOTAL1 lenses evaluated in this study.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | DAILIES TOTAL1
Number analyzed (Participants) | 96
Number analyzed (eyes) | 192
eyes
  20/15 | 95
  20/20 | 92
  20/25 | 5

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, up to approximately 6 to 8 days of contact lens wear.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to DAILIES TOTAL1 lenses evaluated in this study. The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more reporting group.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to delefilcon A contact lenses.
- DAILIES TOTAL1 Ocular; DAILIES TOTAL1 Nonocular: Events reported in this group occurred while exposed to delefilcon A contact lenses.
Arm/Group | Pretreatment | DAILIES TOTAL1 Ocular | DAILIES TOTAL1 Nonocular
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/192 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/192 | 0/96
Other Adverse Events (participants affected / at risk) | 0/96 | 0/192 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study

DOCUMENTS (2):
  • Study Protocol (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT06044948/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT06044948/SAP_001.pdf